CLINICAL TRIAL: NCT04978012
Title: A Phase II Single-site the Study of the Efficacy and Safety of Fluzoparib and Camrelizumab in Treating Patients With Recurrent/Metastatic Nasopharyngeal Carcinoma That Progressed After First-line Chemotherapy
Brief Title: Fluzoparib and Camrelizumab in Treating Patients With R/M NPC That Progressed After First-line Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chaosu Hu, M.D., Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-PAPRi 1.0
Record Dates: First submitted 2021-07-25; First posted 2021-07-27 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Nasopharyngeal Carcinoma; Nasopharyngeal Cancer
Keywords: PARP inhibitor; Fluzoparib; checkpoint inhibitor; PD-1 inhibitor; Camrelizumab
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms | interventions — fluzoparib; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination of Fluzoparib and Camrelizumab (Experimental): Fluzoparib,150mg bid po, d1-21, q3w Camrelizumab 200mg iv, d1, q3w
  Interventions: Drug: Fluzoparib and Camrelizumab

INTERVENTIONS:
Drug: Fluzoparib and Camrelizumab — Maintenance therapy of Fluzoparib and Camrelizumab, until disease progression or intolerable adverse effect.

SUMMARY:
The aim of this study is to define the efficacy and safety of Fluzoparib and Camrelizumab in treating patients with recurrent/metastatic nasopharyngeal carcinoma that progressed after first-line chemotherapy.

DETAILED DESCRIPTION:
Currently, the standard first-line treatment for recurrent/metastatic nasopharyngeal carcinoma is cisplatin-based chemotherapy. The recommended subsequent line therapy is single-agent chemotherapy or single-agent PD-1 antibody (nivolumab or pembrolizumab), according to NCCN guidelines (head and neck cancer, version 2021.3). However, the efficacy of nivolumab or pembrolizumab in subsequent line setting is limited, range from 20-30%. In order to improve the efficacy, we launch this study to evaluate whether combination treatment of PARP inhibitor (Fluzoparib) and PD-1 antibody (Camrelizumab) has the potential to increase efficacy in the subsequent line treatment, meanwhile has tolerable adverse effect.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an informed consent;
2. Age older than 18 years old and younger than 75 years old;
3. Patients with histologically confirmed recurrent/metastatic nasopharyngeal carcinoma, that progressed after at least first-line chemotherapy, according to RECIST 1.1 criteria;
4. No previous treatment of PD-1/L1 inhibitors, CTLA-4 inhibitors, other checkpoint inhibitors or immune modulation therapy, or PARP inhibitors;
5. At least one lesion that fulfills the criteria of "Evaluable Disease" per RECIST 1.1 Criteria;
6. Anticipated overall survival more than 3 months;
7. Satisfactory performance status: ECOG (Eastern Cooperative Oncology Group) scale 0-2;
8. Normal organ function;
9. HBV DNA<500 IU/mL（or 2500 copies/mL）and HCV RNA negative ;
10. Male and no pregnant female, able to adapt birth control methods during treatment.

Exclusion Criteria:

1. Hypersensitivity to Fluzoparib or Camrelizumab;
2. Symptomatic spinal cord compression, or high-risk to develop pathological fracture that requires urgent surgery or radiation;
3. Necrotic disease, high-risk of massive bleeding;
4. Suffered from malignant tumors, except cervical carcinoma in situ, papillary thyroid carcinoma, or skin cancer (non- melanoma) within five years;
5. Severe, uncontrolled heart disease, such as more than NYHA II heart failure, unstable angina pectoris, myocardial infarction within 1 year prior to signing inform consent, severe arrhythmia that requires urgent intervention;
6. Previous treatment of PD-1/L1 inhibitors, CTLA-4 inhibitors, other checkpoint inhibitors or immune modulation therapy, or PARP inhibitors;
7. Receive vaccine or live vaccine within 28 days prior to signing the informed consent;
8. Still suffered from adverse effect (more than CTCAE grade 1), that results from previous treatment;
9. Severe, uncontrolled infections within 28 days prior to signing inform consent;
10. Active, known or suspected autoimmune disease; Type I Diabetes, hypothyroidism those only need hormone replacement therapy, vitiligo or inactive asthma who don't need systemic therapy can recruit;
11. HIV positive;
12. Diagnosed as active pulmonary tuberculosis within one year before signing inform consent; or diagnosed as active pulmonary tuberculosis more than one year, but did not receive standardized anti-tuberculosis treatment;
13. Hepatitis B surface antigen (HBsAg) positive and HBV-DNA ≥500IU/ml, or 2500cps/ml; Positive HCV RNA;
14. History of drug abuse, drug taking, alcohol abuse;
15. Other diseases which may influence the safety or compliance of the clinical trial, such as mental illness, or their family and society factors;
16. Women of child-bearing potential who are pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-07-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Within 2 year post-treatment
  Overall response rate, evaluated by independent radiology review board, according to RECIST 1.1 Criteria

SECONDARY OUTCOMES:
Disease control rate | Within 2 year post-treatment
  Disease control rate, evaluated by independent radiology review board, according to RECIST 1.1 Criteria
Duration of response | Within 2 year post-treatment
  Duration of response, evaluated by independent radiology review board, according to RECIST 1.1 Criteria
Progression-free survival rate at 6 month post-treatment | 6 month post-treatment
  Progression-free survival rate at 6 month post-treatment
Overall survival rate at 6 month post-treatment | 6 month post-treatment
  Overall survival rate at 6 month post-treatment
Progression-free survival rate at 12 month post-treatment | 12 month post-treatment
  Progression-free survival rate at 12 month post-treatment
Overall survival rate at 12 month post-treatment | 12 month post-treatment
  Overall survival rate at 12 month post-treatment
Median progression-free survival | Within 2 year post-treatment
  Median progression-free survival
Median overall survival | Within 2 year post-treatment
  Median overall survival
Adverse effect | Within 2 year post-treatment
  Adverse effect, according to CTCAE 4.0.03 criteria
Overall response rate by different PD-L1 TPS subgroups | Within 2 year post-treatment
  Overall response rate by different PD-L1 TPS subgroups (≥1% vs. <1%; ≥20% vs. <20%; ≥50% vs. <50%）)
Overall response rate by different homologous recombination repair status (HRR) | Within 2 year post-treatment
  Overall response rate by different homologous recombination repair status(germline BRCA mutation/wildtype, HRD positive/negative, germline HRR genes mutations status)

CONTACTS AND LOCATIONS:
Overall Officials: Chaosu Hu, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan Universtiy Shanghai Cancer Centre, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang FH, Wei XL, Feng J, Li Q, Xu N, Hu XC, Liao W, Jiang Y, Lin XY, Zhang QY, Yuan XL, Huang HX, Chen Y, Dai GH, Shi JH, Shen L, Yang SJ, Shu YQ, Liu YP, Wang W, Wu H, Feng H, Yao S, Xu RH. Efficacy, Safety, and Correlative Biomarkers of Toripalimab in Previously Treated Recurrent or Metastatic Nasopharyngeal Carcinoma: A Phase II Clinical Trial (POLARIS-02). J Clin Oncol. 2021 Mar 1;39(7):704-712. doi: 10.1200/JCO.20.02712. Epub 2021 Jan 25. PMID 33492986
- [Background] Ma BBY, Lim WT, Goh BC, Hui EP, Lo KW, Pettinger A, Foster NR, Riess JW, Agulnik M, Chang AYC, Chopra A, Kish JA, Chung CH, Adkins DR, Cullen KJ, Gitlitz BJ, Lim DW, To KF, Chan KCA, Lo YMD, King AD, Erlichman C, Yin J, Costello BA, Chan ATC. Antitumor Activity of Nivolumab in Recurrent and Metastatic Nasopharyngeal Carcinoma: An International, Multicenter Study of the Mayo Clinic Phase 2 Consortium (NCI-9742). J Clin Oncol. 2018 May 10;36(14):1412-1418. doi: 10.1200/JCO.2017.77.0388. Epub 2018 Mar 27. PMID 29584545
- [Background] Lung RW, Hau PM, Yu KH, Yip KY, Tong JH, Chak WP, Chan AW, Lam KH, Lo AK, Tin EK, Chau SL, Pang JC, Kwan JS, Busson P, Young LS, Yap LF, Tsao SW, To KF, Lo KW. EBV-encoded miRNAs target ATM-mediated response in nasopharyngeal carcinoma. J Pathol. 2018 Apr;244(4):394-407. doi: 10.1002/path.5018. Epub 2018 Feb 16. PMID 29230817
- [Background] Tatfi M, Hermine O, Suarez F. Epstein-Barr Virus (EBV)-Related Lymphoproliferative Disorders in Ataxia Telangiectasia: Does ATM Regulate EBV Life Cycle? Front Immunol. 2019 Jan 4;9:3060. doi: 10.3389/fimmu.2018.03060. eCollection 2018. PMID 30662441